CLINICAL TRIAL: NCT05764824
Title: Long-term Effects of Blueberry Supplementation on Brain Health in Older Adults: a Randomized Placebo-controlled Trial
Brief Title: Long-term Effects of Blueberry Supplementation on Brain Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Luc Djousse, MD, ScD, MPH, Lead Investigator and Director of Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022P002554
Record Dates: First submitted 2023-01-31; First posted 2023-03-13 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Decline; Nutrition, Healthy; Brain Injuries
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry group (Active Comparator): Blueberry arm
  Interventions: Dietary Supplement: Blueberry powder
- Control group (Placebo Comparator): Control arm
  Interventions: Other: Controlled and matched powder

INTERVENTIONS:
Dietary Supplement: Blueberry powder — 20 g per day of blueberry powder
  Arms: Blueberry group
Other: Controlled and matched powder — 20 g per day
  Arms: Control group

SUMMARY:
This study will test whether consuming blueberry powder 20g/d for 24 weeks can improve memory and other cognitive function and alter serum biomarkers of brain injury among older adults.

DETAILED DESCRIPTION:
In a randomized, double-blind placebo, controlled design, the investigators will test the effects of 20 g/d of blueberry powder for 24 weeks on cognitive function and serum biomarkers of brain injury among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65-99 years
* Able to travel to Brigham and Women's Hospital for 4 clinic visits

Exclusion Criteria:

* Known allergies to blueberries
* Unable to abstain from blueberry consumption during the study period
* Inability to provide informed consent
* Planned major surgery during study period or recent major surgery up to 3 months before recruitment
* Organ transplant
* Plan to move out of greater Boston area during the study period
* Diagnosis of dementia, severe cognitive decline, end-stage renal disease, substance abuse, insulin-dependent diabetes mellitus, major cancer excluding non-melanoma skin cancer, and schizophrenia.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of neurofilament light (NFL) between baseline and 24 weeks | Baseline and at 24 weeks after the intervention
  Change will be calculated as difference between plasma NFL concentration measured at 24 weeks and NFL concentration measured at baseline.
Change in plasma concentration of phosphorylated tau (pTau-181) between baseline and 24 weeks | Baseline and at 24 weeks post intervention
  Change will be calculated as difference between plasma pTau-181 concentration measured at 24 weeks and plasma concentration of pTau-181 measured at baseline

SECONDARY OUTCOMES:
Change in plasma concentration of glial fibrillary acid protein (GFAB) between baseline and 24 weeks | Baseline and at 24 weeks post intervention
  Change will be calculated as difference between plasma concentration of GFAB measured at 24 weeks and plasma GFAB concentration measured at baseline
Change in concentration of serum non-esterified fatty acids (NEFA) between baseline and 24 weeks | Baseline and 24 weeks post intervention
  Change will be computed as difference between serum concentration of NEFA measured at 24 weeks and serum NEFA concentration measured at baseline
Change in cognitive battery test score between baseline and 24 weeks post intervention | Baseline and at 24 weeks post intervention
  The investigators will use CANTAB (computer-based and interactive software) to complete 8 cognitive battery tests including a) Motor screening task; b) Reaction time; c) Paired associates learning; d) Spatial working memory; e) Pattern recognition memory; f) Delayed matching to sample; g) Rapid visual information processing; and h) Match to sample visual search. The computer automatically calculates a composite score from these 8 tests (a-h) and the investigators will define change in cognitive battery test score as difference in composite score between 24 weeks and baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No